CLINICAL TRIAL: NCT04362332
Title: An Open Label Cluster Randomized Controlled Trial of Chloroquine, Hydroxychloroquine or Only Supportive Care in Patients AdmItted With Moderate to Severe COVID-19
Brief Title: Chloroquine, Hydroxychloroquine or Only Supportive Care in Patients AdmItted With Moderate to Severe COVID-19
Acronym: ARCHAIC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Currently, almost no patients admitted to Dutch hospitals. If any effect of HCQ is to be expected we need more than 1000 inclusions
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Andy I.M. Hoepelman, Head of Infectious Diseases, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL73529.041.20 versie 3
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: chloroquine; hydroxychloroquine; randomized
MeSH Terms: conditions — COVID-19 | interventions — Chloroquine; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: 1. Supportive care + chloroquine base arm: loading dose 600mg, followed by 300mg 12 hours later, followed by 300mg bid for 4 days; total treatment duration of 5 days
  2. Supportive care + hydroxychloroquine arm: loading dose 400mg bid, followed by 200mg bid for 4 days; total treatment duration of 5 days.
  3. Supportive care only.
Masking Description: cluster randomized design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- chloroquine (Active Comparator): 1. Supportive care + chloroquine base arm: loading dose 600mg, followed by 300mg 12 hours later, followed by 300mg bid for 4 days; total treatment duration of 5 days
  Interventions: Drug: Chloroquine Sulfate; Other: Standard supportive care
- hydroxychloroquine (Active Comparator): 2. Supportive care + hydroxychloroquine arm: loading dose 400mg bid, followed by 200mg bid for 4 days; total treatment duration of 5 days.
  Interventions: Drug: Hydroxychloroquine; Other: Standard supportive care
- Supportive care only (No Intervention): 3. Supportive care only.

INTERVENTIONS:
Drug: Chloroquine Sulfate — cluster randomized
  Arms: chloroquine
Drug: Hydroxychloroquine — cluster randomized
  Arms: hydroxychloroquine
Other: Standard supportive care — cluster randomized
  Arms: chloroquine; hydroxychloroquine

SUMMARY:
Rationale: Currently there are no approved treatments for COVID-19. In the Dutch treatment protocol guideline (SWAB) designated treatment is supportive care with the option to add chloroquine base (CQ) or hydroxychloroquine (HCQ). CQ and HCQ are implemented because of their in vitro activity, results from small animal studies, and anecdotal patient's data. There are no published randomized studies with these medications in patients with disease caused by any coronavirus.

Objective: To evaluate if treatment with only supportive care or addition of one of two anti-COVID_19 agents (chloroquine or hydroxychloroquine) results in less disease progression in patients with moderate to severe COVID-19 who require hospital admission.

Study design: Multicentre, cluster randomized cross-over, open label trial. Hospitals will be randomly allocated to one of 3 treatment arms in sequential periods of one week: chloroquine base versus hydroxychloroquine versus supportive care without any drug presumed active against SARS-COV-2. Patients will be treated based on the date of inclusion.

Study population: Adults aged of 18 years and older with moderate to severe, with a NEWS-2 score ≤ 5, laboratory confirmed COVID-19, who require hospital admission in a ward outside the Medium Care or Intensive Care.

Intervention (if applicable): Depending on the treatment arm, the study subject will receive only supportive care or an addition with one of the two agents active against SARS-CoV-2 (chloroquine or hydroxychloroquine).

Main study parameters/endpoints: Disease progression defined as a NEWS-2 score ≥ 7 within 14 days, or admission to Medium Care or Intensive Care Unit, or death.

DETAILED DESCRIPTION:
Study rationale CQ and HCQ were both employed in the treatment of COVID-19 in China. Based on unpublished anecdotal positive results in China, CQ is now implemented in China and the Netherlands in severe COVID-19. HCQ is an analog of CQ with more anti-viral effectivity ex vivo, better safety and tolerability profile.

Rationale for the employment of CQ and HCQ in China comes from the fact that both reduce COVID-19 replication ex-vivo. On top of this, both drugs have clear immunomodulating effects (which is used for various indications to treat rheumatologic diseases) and have shown promising results in patients with dengue and HIV.

Currently, in the Dutch guidelines, for moderate severely ill patients CQ base is the first line of therapy for patients admitted in hospital with moderate to severe COVID-19.

The time needed to "load" the body when using CQ and thus the possible late onset of action suggests that initiation of treatment should be timely. Moreover, the hypothesized mode of action suggests that both HCQ and CQ inhibit cellular replication of COVID-19 but do not have an intrinsic effect on the virus, thus could be best employed when the viral load is low (i.e. early phase of the disease) and thus safe time to improve the subsequent immune response. This underlines that both drugs should be implemented early rather than late in the course of SARS-COV-2 infection.

The investigators propose a cluster randomized controlled study evaluating the value of chloroquine and hydroxychloroquine compared to no antiviral therapy in admitted patients with moderate to severe COVID-19.

Study design:

Population Adult patients with confirmed COVID-19, with moderate to severe symptoms and admitted to the hospital and a NEWS-2 score ≤ 5, will be available for the study.

Intervention

All three treatment arms contain standard supportive care during hospital admission with in two arms an addition with either chloroquine (CQ) or hydroxychloroquine (HCQ) Despite the inclusion of CQ and HCQ as possible additional treatment for COVID-19 in the Dutch treatment guideline, there's no conclusion on the best treatment strategy in this population. Based on pharmacokinetic modelling, and the safety profile, HCQ seems to be more promising than CQ, but both drugs have to be studied in relation to COVID-19. Furthermore, the availability of both drugs might differ from country to country; in the Netherlands for instance, chloroquine is widely available. Therefore, a 1:1:1 trial including standard supportive care with in addition CQ or HCQ as suggested in the LCI/SWAB guideline, the optimal dosages in the different treatment arms are as follows:

1. Supportive care + chloroquine base arm: loading dose 600mg, followed by 300mg 12 hours later, followed by 300mg bid for 4 days; total treatment duration of 5 days
2. Supportive care + hydroxychloroquine arm: loading dose 400mg bid, followed by 200mg bid for 4 days; total treatment duration of 5 days.
3. Supportive care only. Dosage of chloroquine and Hydroxychloroquine will be adjusted, if the patients has a renal impairment with an estimated glomerular filtration rate (eGDR) <10, to 50% of the initial dosage.

If patient will be discharged from hospital before the end of the treatment, treatment is continued outside of the hospital. The general practitioner will receive note of the treatment at discharge.

Main studyendpoint Composite endpoint with disease progression defined as a NEWS2score ≥ 7 within 14 days or resulting in admission to Intensive/Medium Care unit or resulting in death within 14 days.

ELIGIBILITY:
Inclusion Criteria:

* - Patients (≥18 years of age) admitted to the hospital with confirmed COVID-19 and not needing admission to MC or ICU
* Patient has moderate to severe COVID-19. This will be defined as patients with NEWS-2 score ≤ 5.
* Willing and able to give written informed consent

Exclusion Criteria:

* - Severe Covid-19 defined as NEWS-2 score >5 or admission to the ICU needing ventilation or pressure support.
* Contra-indications for hydroxychloroquine or chloroquine
* Unable to take oral medication (chloroquine and hydroxychloroquine can be administered through tube feeding which is considered oral administration)
* Identified allergies to 4-aminoquinoline
* Severe diseases of the blood system
* 6-phosphate dehydrogenase deficiency
* History of acute myocardial infarction, unstable angina pectoris, severe arrhythmia (frequent ventricular, ventricular tachycardia, ventricular fibrillation) in recent 6 months; New York Heart Association (NYHA) level III-IV
* Known corrected QT interval (QTc) ≥ 500ms.
* Uncorrected severe hypokalaemia (< 2,5 mmol/l) or uncorrected severe hypomagnesemia (< 0.6 mmol/l)
* Pancreatitis
* Refusal to participate expressed by patient or legally authorized representative if they are present

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Composite endpoint with disease progression defined as a NEWS2score ≥ 7 within 14 days or resulting in admission to Intensive/Medium Care unit or resulting in death within 14 days. | 14 days
  Composite endpoint with disease progression defined as a NEWS2score ≥ 7 within 14 days or resulting in admission to Intensive/Medium Care unit or resulting in death within 14 days.

SECONDARY OUTCOMES:
Side effects | 28 days
  Secondary study parameters/endpoints Side effects of different drugs leading to regimen change or discontinuation of the antiviral treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UMCU, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months